CLINICAL TRIAL: NCT03658850
Title: Safety and Efficacy of Hydrochlorothiazide in the Treatment of Hypernatremia in Critically Ill Patients: a Randomized Controlled Trial
Brief Title: Safety and Efficacy of Hydrochlorothiazide in the Treatment of Hypernatremia in Critically Ill Patients
Acronym: HYDRA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, André Luiz Nunes Gobatto, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2.603.927
Record Dates: First submitted 2018-05-22; First posted 2018-09-05 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Hypernatremia; Critical Illness
Keywords: hypernatremia; Critical care
MeSH Terms: conditions — Hypernatremia; Critical Illness | interventions — Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): the experimental group will receive one tablet of hydrochlorothiazide in the presentation of 50mg or equivalent enteral solution every 12h (total of 100mg per day) enterally for 3 days.
  Interventions: Drug: Hydrochlorothiazide 50Mg
- Control (Placebo Comparator): placebo group will receive one tablet or equivalent volume of enteral solution of inert substance
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Hydrochlorothiazide 50Mg — for the experimental group received a hydrochlorothiazide tablet on presentation of 50mg or equivalent enteral solution every 12h (total of 100mg per day) enterally on day 0 (D0) until day 3
  Arms: Intervention
Drug: Placebos — for the placebo group will receive one tablet or equivalent volume of enteral solution of inert substance, identical to the hydrochlorothiazide presentations, every 12 hours until day 3
  Arms: Control

SUMMARY:
HYDRA is a randomized clinical trial designed to evaluate safety and efficiency of hydrochlorothiazide in critical patients with hypernatremia

ELIGIBILITY:
Inclusion Criteria:

* hospitalized for intensive care,
* Over 18 years of age,
* Two serum sodium measurements above 145 mEq / L (with no pre-determined interval between them),
* Mean arterial pressure greater than 65mmHg

Exclusion Criteria:

* Absence of consent to participate in the study
* Cardiac index below 2.5L / min / m2 OR signs of ineffective circulation (capillary filling time greater than 2 seconds, cold or sticky skin) OR arterial lactate> 4mMol / L.
* Use of vasopressors at doses greater than 0.1 mcg / kg / min of noradrenaline or with initiation or increase of dose within less than one hour before inclusion in the study.
* Unavailable enteral route.
* Use of hydrochlorothiazide in the last 7 days of ICU admission.
* History of allergy or intolerance to hydrochlorothiazide or other thiazides.
* Nephrogenic Diabetes Insipidus.
* Renal impairment KDIGO 3
* Indication of renal replacement therapy.
* Acute neurological insult.
* Heart failure American Heart Association classification (AHA), class D.
* Liver cirrhosis Child-Pugh C.
* Pregnant women
* Exclusive palliative care
* Dying, with expected survival less than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-10 (Estimated); Study Completion 2020-03-10 (Estimated)

PRIMARY OUTCOMES:
hypernatremia correction | DAY 3
  proportion of patients with hypernatremia correction (serum sodium below 145 mEq / L) at the end of Day 3

SECONDARY OUTCOMES:
renal replacement therapy | 6 months
  need to renal replacement therapy
mechanical ventilation | 6 months
  incidence of mechanical ventilation
vasoactive drugs | 6 months
  need for vasoactive drugs
mortality | 6 months
  hospital mortality
serious adverse events | 6 months
  incidence of serious adverse events 37/5000 incidence of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: André LN Gobatto, p.h.d, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil